CLINICAL TRIAL: NCT00255242
Title: Effect of Simvastatin on CF Airway Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Nathan Kraynack, MD, Akron Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRAYNA04A0; KRAYNA04A0
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2008-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Airway Inflammation; Cytokines; Simvastatin; HMG-CoA reductase inhibitors; Rho GTP-ase
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Simvastatin treatment for 28 days — 40 mg / day

SUMMARY:
Individuals with cystic fibrosis (CF) have persistent infection in the airways, which the body attempts to fight by recruiting immune cells (neutrophils) to the lung. The immune system and neutrophils are unable to completely kill the bacteria, and the response to the infection leads to inflammation (swelling) of the airways and lung damage. Nitric oxide (NO) has anti-bacterial and anti-inflammatory properties in the lung. NO production is decreased in CF patients, and may contribute to the persistent infection and inflammation. Increasing the production of NO in the airways of CF patients may help decrease this inflammation and infection.

Rho GTPases are molecules in the cells that line the airways that decrease the protein that makes nitric oxide (NOS). Rho proteins also increase inflammation in these cells. Rho proteins are increased in CF cells, and may partially explain the low NO and high inflammation seen in CF. Blocking the Rho protein in CF cells increases NOS, which can then produce more NO. The Rho protein can be inhibited with a drug, simvastatin (Zocor®). Simvastatin is used by millions of people to lower their cholesterol, is very safe, has few side-effects and is approved for use in children greater than 10 years of age. We propose that treating CF patients with simvastatin will increase NO produced (exhaled NO), and may decrease airway inflammation.

If simvastatin has these expected effects in CF, it would be another drug that has potential to become a new therapy to fight the debilitating lung damage of the disease.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) lung disease is characterized by chronic bacterial infection and excessive inflammation. The airways of patients with CF contain large amounts of neutrophils, neutrophil products, and pro-inflammatory mediators. This inflammatory response may be linked to the loss of CFTR function. It is unknown, however, what signaling mechanisms link a loss of CFTR function to the excessive inflammatory response. Several signaling pathways are dysregulated in CF epithelial cells. Among these is the pathway that leads to the production of nitric oxide (NO). Reduced production of NO, which has important antibacterial and anti-inflammatory effects in the airway, may contribute to the establishment of the chronic bacterial infection and the development of the subsequent overzealous inflammatory response in CF.

NO synthesis in the airway epithelium is regulated by nitric oxide synthase 2 (NOS2). NOS2 expression is negatively regulated by the Rho GTPases, which are over-expressed in CF and may also play a role in the inflammatory dysregulation characteristic of the lung disease. Inhibition of the Rho GTPases with 3-hydroxy-3-methylglutaryl-CoA reductase (HMG-CoAR) inhibitors, such as simvastatin (Zocor®), increases NOS2 protein expression in CF airway epithelial cells. The statins have also been shown to have potent systemic anti-inflammatory effects, many of which may be pertinent to CF. We propose to test the hypothesis that HMG-CoAR inhibitors, such as simvastatin, have the potential to correct abnormalities in NO production and decrease inflammation in the airways of patients with CF. The following specific aims will be pursued in this application: 1) To determine the effect of simvastatin treatment on exhaled nitric oxide (eNO) concentrations in subjects with CF; 2) To determine the effect of simvastatin treatment on inflammation and NOS2 production in the airway of subjects with CF, as determined by quantitative RT-PCR for IL-6, IL-8, and NOS2 mRNA in nasal epithelial cells; 3) To determine if quantitative RT-PCR measurements on nasal epithelial cells might be used as a surrogate marker of lower airway inflammation by comparing the measures obtained from nasal epithelial scrapes with inflammatory measurements obtained from induced sputum.

This study has the potential to identify a new agent that targets a signaling pathway (Rho GTPase) that appears to be dysregulated in CF, and thus, may exert multiple beneficial effects in the CF airway including increasing airway NO concentrations, decreasing neutrophil influx and reducing production of inflammatory mediators. In addition to evaluating the anti-inflammatory effects of statins in CF, this study presents an opportunity to evaluate alternative outcome measures of CF airway inflammation. The results of this study will provide important information regarding the feasibility of using nasal epithelial sampling as a relatively non-invasive measure of airway inflammation in CF.

ELIGIBILITY:
Inclusion Criteria:

* Cystic Fibrosis
* > 9 yrs of age
* Clinically stable
* FEV1 > 50% predicted

Exclusion Criteria:

* Hepatic disease
* B. cepacia
* corticosteroids
* symptomatic allergic rhinitis

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-07; Primary Completion 2008-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Specific Aim 1: To determine the effect of simvastatin treatment on exhaled NO, eNO measurements from the Run-in phase will be compared to the Treatment phase. | 1 month

SECONDARY OUTCOMES:
Specific Aim 2: Synthesis of the following markers will be measured in nasal epithelial samples by quantitative PCR. | 1 months
Specific Aim 3: Cell and differential counts will be obtained in induced sputum as an overall measure of the inflammatory response.Concentrations of neutrophil products (elastase) and cytokines also will be measured in induced sputum. | 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathan C Kraynack, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States